CLINICAL TRIAL: NCT04517708
Title: Effectiveness of Nutritional Interventions for Cancer Patients Undergoing Chemotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hanoi Medical University (Other)
Collaborators: Ministry of Health of Vietnam (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 187/HĐĐĐĐHYHN
Record Dates: First submitted 2020-08-14; First posted 2020-08-18 (Actual); Last update posted 2020-08-18 (Actual); Status verified 2020-08

CONDITIONS: Gastric Cancer; Colon Cancer
MeSH Terms: conditions — Stomach Neoplasms; Colonic Neoplasms | interventions — Nutrition Assessment

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Regarding the intervention group, patients were treated with the intervention regimen, which consisted of:
  * Nutritional counseling
  * Each patient was assigned a specific menu which were prepared by research members during the time of staying at the hospital. Before discharge, patients were instructed on preparing their diets at home with the recommended amount of energy and protein and given formula milk within two months.
  Interventions: Other: Nutritional counseling
- Control group (No Intervention): Patients had diets based on their demands

INTERVENTIONS:
Other: Nutritional counseling — Each patient was assigned a specific menu which were prepared by research members during the time of staying at the hospital. Before discharge, patients were instructed on preparing their diets at home with the recommended amount of energy and protein and given formula milk within two months
  Arms: Intervention group

SUMMARY:
This study aims to estimate the effects of nutritional interventions on the improvement of nutritional status and quality of life (QoL) among gastrointestinal patients in Vietnam

DETAILED DESCRIPTION:
A quasi-experiment with intervention and control groups for pre- and post-intervention assessment was carried out at the Department of Oncology and Palliative Care - Medical University Hospital from 2016 to 2019. 60 gastrointestinal cancer patients were recruited in each group. At stage 1, we selected patients of the intervention group who met the inclusion criteria to receive nutritional counseling and diet at the hospital. At stage 2, we chose patients who were eligible but did not accept the nutritional counseling and diet at the hospital. Participants in both groups were paired together according to the following criteria: 1) Age group: <40 years old, 40-65 years old and >65 years old; 2) Gender: Male and female; 3) Types of cancer: stomach cancer and colon cancer; 4) Disease stages: stage 1-2 and stage 3-4.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 years old or above
* diagnosed with stomach or colon cancer;
* at the initial of receiving chemotherapy treatment;
* indicated for oral feeding;
* not having co-morbidities of chronic diseases such as kidney failure, heart failure, liver failure, diabetes;
* having ability to communicate with data collectors and both attending doctors and agreeing to involve in the study

Exclusion Criteria:

* treated by other methods such as radiation, endocrine, immunity;
* undergoing terminal palliative care;
* having contraindications to oral feeding/enteral nutrition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2016-01-15 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-12-15 (Actual)

PRIMARY OUTCOMES:
Change of nutritional status after 8 weeks | Baseline and 8 weeks
  The Scored Patient-Generated Subjective Global Assessment (PG-SGA) was used as the preeminent interdisciplinary patient assessment among patients with oncology. This tool includes (1) four patient-generated historical components (Weight History, Food Intake, Symptoms, Activities and Function); (2) the professional part (Diagnosis, Metabolic stress, and Physical Exam); (3) the Global Assessment (A = well-nourished, B = moderately malnourished, C = severely malnourished); (4) the total score, and nutritional triage recommendations. Changes in anthropometric indicators were also reported (weight, MUAC, muscle mass)
Change of quality of life after 8 weeks: European Organisation for Research and Treatment of Cancer (EORTC) version 3.0 | Baseline and 8 weeks
  We utilized the European Organisation for Research and Treatment of Cancer (EORTC) version 3.0, which is an integrated and modular approach to holistically evaluate the QoL of patients with cancer.all dimensions of the tool will range from 0 to 100, in which a higher score presents a better level of functioning/the global health status or a worse level of symptoms.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nguyen LT, Dang AK, Duong PT, Phan HBT, Pham CTT, Nguyen ATL, Le HT. Nutrition intervention is beneficial to the quality of life of patients with gastrointestinal cancer undergoing chemotherapy in Vietnam. Cancer Med. 2021 Mar;10(5):1668-1680. doi: 10.1002/cam4.3766. Epub 2021 Feb 7. PMID 33550719